CLINICAL TRIAL: NCT03609671
Title: A Pilot Study: Emotions Immunology and Breast Cancer
Brief Title: Emotions Immunology and Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Luz A. Venta, MD (Other)
Responsible Party: Sponsor-Investigator, Luz A. Venta, MD, Principal Investigator, Houston Methodist Hospital Physician, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00013603
Record Dates: First submitted 2018-07-24; First posted 2018-08-01 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer; Triple Negative Breast Cancer; Emotions; Immunology
Keywords: Breast Cancer; Emotions Immunology
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to two groups.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care + Intervention (Individualized Therapy) (Experimental): Intervention (individualized therapy) plus Standard of Care, and the completion of a psychological questionnaire at chemotherapy start and at the end, approximately four to six months later.
  Interventions: Behavioral: Standard of Care + Experimental Individualized Therapy
- Control Group: Standard of Care (Other): Standard of Care plus the completion of a psychological questionnaire at the beginning of the chemotherapy and at the end, approximately four to six months later.
  Interventions: Other: Control: Standard of Care

INTERVENTIONS:
Behavioral: Standard of Care + Experimental Individualized Therapy — Participants will receive standard of care plus supportive psychotherapy for a one hour, weekly, during the time they are undergoing neoadjuvant treatments.
  Other Names: Individualized Therapy
  Arms: Standard of Care + Intervention (Individualized Therapy)
Other: Control: Standard of Care — Participants will undergo standard of care only (no Intervention/no individualized therapy) .
  Other Names: No intervention; No Individualized Therapy
  Arms: Control Group: Standard of Care

SUMMARY:
Pilot study representing a proof of concept regarding the potential for immune system enhancement with psychotherapy, resulting in improved immunological response at lumpectomy or mastectomy in patients undergoing neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Study participants will receive be randomized to the experimental group (receive individualized psychotherapy + standard of care) or the control group (standard of care) and both groups will complete psychological questionnaires. Both groups will have blood sampling and have their biopsied tissue read for immunological factors.

Patients with triple negative breast cancer or with breast cancers presenting at a large size (greater than one centimeter) have a worst prognosis than other types of breast cancer or cancers that are diagnosed when smaller than one centimeter. For these patients, neoadjuvant chemotherapy, that is chemotherapy given before surgical removal of the cancer, is often used. Common indications for using neoadjuvant therapy include: available clinical trial, learning about the tumor response in vivo to a particular chemotherapy and shrinking the tumor so as to convert a mastectomy to a lumpectomy at the time of resection. In patients receiving neoadjuvant treatment, there is usually 6-months between the diagnosis and the surgical breast tumor resection during which the chemotherapy is administered, and during that time patients are offered support group therapy. Although the prognosis for breast cancer patients has improved, this subset of patients still poses a clinical challenge.

Growing evidence in the psychological field has documented a link between the immune system and psychological factors, emphasizing that stress and trauma are detrimental to the ability and effectiveness of the immune system and emphasizing that mental health has an importance not only in and of itself on how the person feels, but also translates into physical health at least in part through the immune system. Personality traits and other emotional factors remain as viable candidates contributing to the development of malignancies, but the research in this area is confusing. For example, many authors report that depressed women are more prone to develop breast cancer than others, while other research has failed to find such a connection.

Nevertheless, many clinicians notice that cancer tends to present after a major loss or emotional trauma. Some research suggests that the suppression of negative emotions or difficulty expressing emotions such as anger and hostility are characteristic of the cancer-prone personality, so that in a typical study, clinicians who interviewed patients prior to breast biopsy were able to predict the presence of a malignancy in 94% of cases based on psychological factors alone. Similarly, a study has been able to predict with 75% accuracy those patients who had early cancer with no knowledge of their Pap smear results, based on the presence of extreme hopelessness. However, although there are many similar studies, other researchers have not been able to confirm the importance of emotional factors.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant adult (eighteen years old or older) women with a diagnosis of breast cancer
* Planned to receive neoadjuvant chemotherapy for about six month duration
* Must be fluent in speaking, reading and writing English
* Not planning on undergoing individual psychotherapy during the study time outside the study.
* Biopsy procedure to be performed with surgical treatment planned at Houston Methodist System

Exclusion Criteria:

* Pregnant or planned to become pregnant
* Patient not fluent in English
* Patients undergoing individual psychotherapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Questionnaire#1, Adverse Childhood Experience (ACE). | Baseline pre-chemotherapy and post-chemotherapy (about 4-6 months later).
  The self-reported Adverse Childhood Experience Questionnaire measures different types of abuse, neglect, and other hallmarks of a challenging childhood. Scores range from 0-10, with 10 indicating highest childhood abuse &/or neglect exposure with greater risk for negative consequences later in life, and 0 is lowest exposure and lower risk for negative consequences.questionnaires with immune responses. Pathologic tumor response is our measurable endpoint, focusing on immune cells in the tumor bed at lumpectomy or mastectomy.
Questionnaire#2, Depression, Anxiety, and Stress Scale (DASS). | Baseline pre-chemotherapy and post-chemotherapy (about 4-6 months later).
  The self-reported Depression, Anxiety, and Stress Scale Questionnaire is 3-part tool that measures motional states of depression, anxiety, and stress. Scores range from 0-42 for depression, 0-42 for anxiety and 0-42 for stress. A score closer to 42 for each state is indicative of extremely severe symptoms while a score closer to 0 indicates normal to mild symptom scores.
Questionnaire#3, Experiences in Close Relationships-Revised (ECR-R). | Baseline pre-chemotherapy and post-chemotherapy (about 4-6 months later).
  The self-reported Experiences in Close Relationships-Revised Adult Attachment Questionnaire is a tool that measures how an individual behaves in relationships with others. Scores range from 0-5. A score closer to 0 is indicative of attachment while a score closer to 5 indicates signs of attachment-avoidance.
Questionnaire#4, Functional Assessment of Cancer Therapy - Breast Cancer (FACT-B, version 4). | Baseline pre-chemotherapy and post-chemotherapy (about 4-6 months later).
  The self-reported Functional Assessment of Cancer Therapy Questionnaire is a tool that measures how an individual behaves in relationships with others. Scored in a 5 point scale with a total score ranging from 0 to 164, with a higher score indicative of better health related quality of life.
Questionnaire#5, Benefit Finding Scale (BFS). | Baseline pre-chemotherapy and post-chemotherapy (about 4-6 months later).
  The self-reported Benefit Finding Questionnaire is a tool that measures how an individual might feel their cancer diagnosis contributes to their outlook on life. Scored in a 5 point scale with total scores ranging from 17-85. Higher scores indicate more benefit derived from breast cancer.
Questionnaire#6, Acceptance and Action Questionnaire - II (AAQ-II) | Baseline pre-chemotherapy and post-chemotherapy (about 4-6 months later).
  The self-reported Acceptance and Action Questionnaire - II is a tool that measures psychological inflexibility and experiential avoidance. Score in a 7 point scale, range 7 to 49. A higher score indicates greater levels of psychological inflexibility .

CONTACTS AND LOCATIONS:
Overall Officials: Luz A. Venta, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (2):
- United States (2):
  - Houston Methodist Hospital Cancer Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided
to be determined

REFERENCES:
- [Background] [1.] Baumeister, D., et al. Childhood trauma and adult inflammation: a meta-analysis of peripheral C-reactive protein, interleukin-6 and tumor necrosis factor-α. Molecular Psychiatry: 2015: 1-8. [2.] Bleiker, E.M. et al. Personality factors and breast cancer development: a prospective longitudinal study. Journal of the National Cancer Institute; 1996: 1478-1482. [3.] Brod, S., et al. 'As above, so below." Examining the interplay between emotion and the immune system. Immunology, 2014: 143, 311-318. [4.] Buchheim A, Viviani R, Taubner S, et al. EPA-0142 - Neural changes in depressed patients during psychodynamic psychotherapy: An fMRI Study. European Psychiatry [serial online]. January 1, 2014;29(1, Number 1 Supplement 1):1. [5.] Carrig M, Kolden G, Strauman T. Using functional magnetic resonance imaging in psychotherapy research: A brief introduction to concepts, methods and task selection. Quantitative and qualitative methods in psychotherapy research [e-book]. New York, NY, US: Routledge/Taylor & Francis Group; 2014:72-84. [6.] Dumas J, Makarewicz J, Newhouse P, et al. Chemotherapy altered brain functional connectivity in women with breast cancer: a pilot study. Brain Imaging And Behavior [serial online]. December 1, 2013;7(4):524-532. [7.] Spiegel, D. Minding the body: Psychotherapy and cancer survival. British Journal of Health Psychology, 2014, 19: 465-485. [8.] Temoshok L. Personality, coping style, emotion and cancer: towards an integrative model. Cancer Surv 1987:6:545-67. [9.] Wirsching, M., et al., Psychological identification of breast cancer patients before biopsy. Journal of Psychosomatic Research, 1982: 26(1): 1-10. [10.] Zonderman AB, et al. Depression as a risk for cancer morbidity and mortality in a nationally representative sample. JAMA 1989;262:1191-5. [11.] Persky VW, et al. Personality and risk of cancer: 20-year follow-up of the Western Electric Study. Psychosom Med 1987;49:435-49. [12.] Chida, Y., Hamer, M., Wardle, J., & Steptoe, A. (2008). Do stress-related psychosocial factors contribute to cancer incidence and survival?. Nature Clinical Practice. Oncology, 5(8), 466-475. doi:10.1038/ncponc1134 [13.] Fagundes, C. P., Lindgren, M. E., & Kiecolt-Glaser, J. K. (2013). Psychoneuroimmunology and Cancer: Incidence, Progression, and Quality of Life. In Psychological Aspects of Cancer (pp. 1-11). Springer US. [14.] Lillberg, K., Verkasalo, P. K., Kaprio, J., Teppo, L., Helenius, H., & Koskenvuo, M. (2003). Stressful life events and risk of breast cancer in 10,808 women: a cohort study. American Journal Of Epidemiology, 157(5), 415-423. [15.] Lutgendorf, S. K., Johnsen, E. L., Cooper, B., Anderson, B., Sorosky, J. I., Buller, R.E., & Sood, A. K. (2002). Vascular endothelial growth factor and social support in patients with ovarian carcinoma. Cancer, 95(4), 808-815. [16.] Lutgendorf, S. K., Lamkin, D. M., Jennings, N. B., Arevalo, J. G., Penedo, F., DeGeest, K., & ... Sood, A. K. (2008). Biobehavioral influences on matrix metalloproteinase expression in ovarian carcinoma. Clinical Cancer Research: An Official Journal Of The American Association For Cancer Research, 14(21), 6839 6846. doi:10.1158/1078-0432.CCR-08-0230 [17.] Pocock, S.J., & Simon, R. (1975). Sequential Treatment Assigment with Balancing for Prognostic Factors in the Controlled Clinical Trial, Biometrics, 31(1), 103-115. doi.org/10.2307%2F2529712 [18.] Han, B., Enas, N. H. and McEntegart D. (2009). Randomization by minimization for unbalanced treatment allocation. Statistics in Medicine, 28(27), 3329-3346.